CLINICAL TRIAL: NCT03827200
Title: A Phase II, Single-arm, Open-label Study to Characterise the Effect on Portal Pressure, the Effect on Renal Function and the Pharmacokinetic Profile of N-003 in Patients With Decompensated Cirrhosis
Brief Title: A Study Evaluating the Utility of Ambrisentan in Lowering Portal Pressure in Patients With Liver Cirrhosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment, result of COVID-19 pandemic
Sponsor: Noorik Biopharmaceuticals AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-003-CRD003; 2018-002088-25 (EudraCT Number)
Record Dates: First submitted 2019-01-25; First posted 2019-02-01 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Cirrhosis; Portal Hypertension; Ascites
Keywords: Cirrhosis; Portal Hypertension; Ambrisentan; N-003; Hepatic Vein Pressure Gradient; HVPG; Refractory Ascites; Varices, Esophageal; Variceal Hemorrhage; Hepatitis B; Hepatitis C; Non-Alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis; Ascites
MeSH Terms: conditions — Fibrosis; Hypertension, Portal; Ascites; Esophageal and Gastric Varices; Hepatitis B; Hepatitis C; Non-alcoholic Fatty Liver Disease | interventions — ambrisentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ambrisentan (Experimental): Ambrisentan
  Interventions: Drug: Ambrisentan

INTERVENTIONS:
Drug: Ambrisentan — Ambrisentan will be administered subcutaneously at the Hospital on the days of HVPG deterination and taken orally at home between visits.
  Other Names: N-003

SUMMARY:
Endothelin is a human hormone which has been associated with increased portal pressure in patients with liver cirrhosis (also called portal hypertension). Ambrisentan blocks the effects of endothelin. The purpose of this study is to evaluate the effect of ambrisentan on portal pressure and renal function in patients with advanced liver cirrhosis and with portal hypertension. In this study, portal pressure will be determined at multiple times with the aid of a catheter inserted into the body of the patient. The effect of ambrisentan on the function of the kidney will also be investigated. This study will also evaluate the concentrations of ambrisentan in blood in patients with liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent including data protection declaration prior to study participation
* Subjects with confirmed cirrhosis (by biopsy, ultrasound, and/or laboratory examinations)
* Ascites Grade II or Grade III at screening currently treated with at least one diuretic or the subject is considered intolerant to diuretics in the investigator's opinion

Exclusion Criteria:

* Age <18 years of age
* Any of the following laboratory findings at the time of screening

  * Serum creatinine level >1.5mg/dL (>132 µmol/L)
  * Serum Na+ < 125 meq/L
  * Serum K+ ≥ 5.5 meq/L
  * Serum bilirubin ≥ 5 mg/dL (85.5 µmol/L)
  * INR >3.0
* Women of childbearing potential with no effective contraceptive method (women of childbearing potential [pre-menopausal, not surgically sterile for at least 3 months prior to the time of screening] must have a confirmed negative serum β-hCG pregnancy test prior to enrolment and at Baseline Visit. They must use an effective contraceptive method throughout the study, and agree to repeat serum β-hCG pregnancy tests at designated visits)
* Pregnancy or lactation
* Systolic blood pressure <90 mmHg or diastolic blood pressure <60 mmHg
* Sepsis and/or uncontrolled bacterial infection
* Current or recent documented nephrotoxicity (within 4 weeks)
* Hepatic Encephalopathy above grade 1
* History of variceal bleeding in the last 2 months
* Suspicion of active alcohol consumption in the last 3 months
* History of liver or kidney transplantation
* History of Transjugular Intrahepatic Portosystemic Shunt (TIPS)
* Suspected occlusive portal vein or splenic vein thrombosis
* Hepatocellular carcinoma (HCC) beyond the Milan criteria
* Acute Liver Failure or superimposed acute liver injury due to drugs (e.g., acetaminophen), dietary supplements, herbal preparations, viral hepatitis, or toxins
* Severe cardiovascular disease, including, but not limited to, unstable angina, pulmonary oedema, congestive heart failure
* Current or recent (within 30 days) renal replacement therapy (RRT)
* If on beta-blockers, a change in dose or drug within last 15 days prior to screening
* Use of any other endothelin receptor antagonist, octreotide, midodrine, terlipressin in last 15 days prior to screening
* Known hypersensitivity to contrast-media
* Any clinically significant abnormality identified on physical examination, laboratory tests, ECG or vital signs at the time of screening that in the judgment of the investigator or any sub-investigator would preclude safe completion of the study or constrains the assessment of efficacy
* Known sensitivity to ambrisentan or any of the excipients of the formulation
* Participation in other clinical research involving investigational medicinal products within 30 days of enrolment
* Subjects who have difficulties in understanding the language in which the study information is given
* Subjects who do not agree to the transmission of their anonymous data within the liability of documentation and notification
* Staff of the study centre, staff of the sponsor or Clinical Research Organization (CRO), the investigator himself or close relatives of the investigator.

Cardiac and Pulmonary Haemodynamic Study exclusion Criteria: Subjects fulfilling any of the exclusion criteria below may participate in the study, but will not undergo cardiac and pulmonary catheterisation:

* Significant arrhythmias, which include any of the following: sustained ventricular tachycardia, bradycardia with sustained ventricular rate < 45 beats per minute or atrial fibrillation/flutter with sustained ventricular response of > 90 beats per minute at rest, or Long QT syndrome or QTc > 450 ms
* Significant left ventricular outflow tract obstructions (e.g., severe valvular aortic stenosis, obstructive cardiomyopathy), severe mitral stenosis, restrictive amyloid myocardiopathy, acute myocarditis
* Severe aortic insufficiency or severe mitral regurgitation for which surgical or percutaneous intervention is indicated
* Major neurologic event including cerebrovascular events, within 30 days prior to screening
* Clinical evidence of acute coronary syndrome currently or within 30 days prior to screening
* Permanent pacemaker, cardiac resynchronisation device or implantable cardioverter-defibrillator in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Mean change in Hepatic Vein Pressure Gradient (HVPG) from Baseline to Day 14 | 14 Days
  Baseline HVPG is defined as the HVPG assessment performed prior to the first study drug administration. Day 14 HVPG is defined as the HVPG assessment prior to the last dose of study drug. The mean change in HVPG will be calculated as the difference between the HVPG assessment performed at Day 14 and the HVPG assessment performed at baseline

SECONDARY OUTCOMES:
Change in 24-hour Urinary Sodium Volume (UNaV) | 48 hours
  The change in 24-hour Urinary Sodium Volume (UNaV) will be calculated as the difference in 24-hour UNaV at Baseline and the 24-hour UNaV at Day 1 (after the first study drug administration).
  Urinary sodium volume collected in the 24 hours of baseline will be compared to the Urinary sodium volume collected in the 24 hours after the first dose of the drug. Collection of urine will be ongoing for 48 hours in total.
Change in weight | 28 days
  The change in weight will be calculated as the difference in weight at baseline and weight recorded throughout the study
Change in abdominal girth | 28 days
  The change in abdominal girth will be calculated as the difference in abdominal girth at baseline and abdominal girth recorded throughout the study
Change in Model of End-Stage Liver Disease (MELD) score | 28 days
  The change in MELD score will be calculated as the difference in MELD score at baseline and the MELD scores recorded throughout the study.
  The MELD score is calculated according to the following formula:
  MELD = 3.78×ln[serum bilirubin (mg/dL)] + 11.2×ln[INR] + 9.57×ln[serum creatinine (mg/dL)] + 6.43
  The MELD score provides an indication of the anticipated mortality observed in previous studies when subjects were followed for 3-months, according to the following ranges:
  71.3% mortality if score is 40 points or more
  52.6% mortality if score between 30-39 points
  19.6% mortality if score between 20-29 points
  6.0% mortality if score between 10-19 points
  1.9% mortality if score 9 points or less
  The MELD score will be calculated at each visit during a 28 day period.
Change in Child-Pugh score | 28 days
  The change in Child-Pugh score will be calculated as the difference in Child-Pugh score at baseline and the Child-Pugh scores recorded throughout the study
  The Child-Pugh score provides information on the prognosis of a patient based on 5 clinical parameters which are individually graded. These parameters include laboratory values and other clinical information from the patient, such as the presence of ascites or hepatic encephalopathy. A lower score signifies a better chance and a higher score indicates a worse chance of survival at one year. Once the score is calculated it is further subclassified into three stages, depending on the score:
  Child A - the score is between 5 and 6. The survival rate is 100%
  Child B - the score is between 7 and 9. The survival rate is 80%
  Child C - the score is between 10 and 15. The survival rate is 45%
Change in Cardiac Output | 14 days
  The change in Cardiac Output will be calculated as the difference in Cardiac Output at baseline and the Cardiac Output recorded at Day 14
Change in Cardiac Index | 14 days
  The change in Cardiac Index will be calculated as the difference in Cardiac Index at baseline and the Cardiac Index recorded at Day 14
Change in Pulmonary Capillary Wedge Pressure | 14 days
  The change in Pulmonary Capillary Wedge Pressure will be calculated as the difference in Pulmonary Capillary Wedge Pressure at baseline and the Pulmonary Capillary Wedge Pressure recorded at Day 14
Change in Pulmonary Arterial Pressure | 14 days
  The change in Pulmonary Arterial Pressure will be calculated as the difference in Pulmonary Arterial Pressure at baseline and the Pulmonary Arterial Pressure recorded at Day 14
Change in Central Venous Pressure | 14 days
  The change in Central Venous Pressure will be calculated as the difference in Central Venous Pressure at baseline and the Central Venous Pressure recorded at Day 14

OTHER OUTCOMES:
Proportion of patients achieving a 20% reduction in HVPG at Day 14 from baseline | 14 days
Proportion of patients achieving a 10% reduction in HVPG at Day 14 from baseline | 14 days
Proportion of patients achieving an HVPG of 10 mmHg or less at Day 14 from baseline | 14 days
Proportion of patients achieving an HVPG of 12 mmHg or less at Day 14 from baseline | 14 days

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Clinic Barcelona, Barcelona, Catalonia
  - Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda, Madrid
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid